CLINICAL TRIAL: NCT00694382
Title: A Multinational, Randomized, Double Blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of AVE5026 in the Prevention of Venous Thromboembolism (VTE) in Cancer Patients at High Risk for VTE and Who Are Undergoing Chemotherapy
Brief Title: Evaluation of AVE5026 in the Prevention of Venous Thromboembolism in Cancer Patients Undergoing Chemotherapy
Acronym: SAVE-ONCO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EFC6521; 2007-007943-29 (EudraCT Number)
Record Dates: First submitted 2008-05-07; First posted 2008-06-10 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Venous Thromboembolism; Cancer
Keywords: chemotherapy
MeSH Terms: conditions — Venous Thromboembolism; Neoplasms | interventions — AVE 5026

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Semuloparin (Experimental): Semuloparin sodium 20 mg once daily until change in chemotherapy regimen
  Interventions: Drug: Semuloparin sodium
- Placebo (Placebo Comparator): Placebo (for semuloparin) once daily until change in chemotherapy regimen
  Interventions: Drug: Placebo (for semuloparin)

INTERVENTIONS:
Drug: Semuloparin sodium — 0.4 mL solution in ready-to-use 0.5 ml pre-filled syringe
  Subcutaneous injection
  Other Names: AVE5026
  Arms: Semuloparin
Drug: Placebo (for semuloparin) — 0.4 mL solution in ready-to-use 0.5 ml prefilled syringe strictly identical in appearance but without active component
  Subcutaneous injection
  Arms: Placebo

SUMMARY:
The primary objective was to compare the efficacy of once daily subcutaneous injections of Semuloparin sodium (AVE5026) with placebo in the prevention of venous thromboembolism [VTE] in cancer patients at high risk for VTE and who were undergoing chemotherapy.

The secondary objectives were to evaluate the safety of Semuloparin sodium (AVE5026), to document Semuloparin sodium (AVE5026) exposures, to try identifying a metagene predictor of VTE and to assess the survival status at one year in this population.

DETAILED DESCRIPTION:
Randomization had to take place just prior to the first study drug injection (randomization ratio 1:1).

The study period per participant was variable depending on the duration of chemotherapy. It included:

* a screening period up to 3 weeks,
* a double-blind treatment period,
* a follow-up period of 1 month.

Study end date was at the latest 7 months following the randomization of the last participant (6 months treatment and 1 month follow-up).

ELIGIBILITY:
Inclusion Criteria:

Cancer patient with metastatic or locally advanced solid tumor of lung, pancreas, stomach, colon/rectum, bladder or ovary initiating a (new) course of chemotherapy with a minimum intent of 3 months therapy

Exclusion Criteria:

* Required systematic venous thromboprophylaxis or curative treatment with anti-coagulant or thrombolytic;
* High risk of bleeding;
* Severe renal impairment (estimated creatinine clearance <30 mL/min);
* ECOG (Eastern Cooperative Oncology Group) performance status 3 & 4;
* Major surgery within 4 weeks before randomization;
* Known hypersensitivity to unfractionated heparin [UFH] or low molecular weight heparin [LMWH].

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3212 (Actual)
Dates: Start 2008-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Who Experienced Venous Thromboembolism Event [VTE] or VTE-related Death | From randomization up to 3 days after last study drug injection
  VTE included any symptomatic Deep Vein Thrombosis [DVT] of lower or upper limbs and any non-fatal Pulmonary Embolism [PE] as confirmed by a Central Independent Adjudication Committee [CIAC] after review of compression ultrasound or venography for DVT, ventilation/perfusion lung scan, pulmonary angiogram or spiral computer tomography lung scan for PE.
  VTE-related death included fatal PE and unexplained deaths without confirmatory autopsy. Any sudden death could be classified as fatal PE by the CIAC unless diagnostic test results strongly indicated an alternative diagnosis".
Time-to-first Occurrence of VTE or VTE-related Death (Cumulative Incidence Function) | From randomization up to 3 days after last study drug injection
  Participants alive and not having experienced VTE were right censored at last study drug injection plus 3 days. In order to correct for competing risks (Deaths other than VTE-related death), a model of cause-specific hazards was used to estimate the Cumulative incidence Function with Prentice non-parametric estimator.

SECONDARY OUTCOMES:
Percentage of Participants who required the initiation of curative anticoagulant or thrombolytic treatment after VTE assessment | From randomization up to 3 days after last study drug injection
  Initiation of curative anticoagulant or thrombolytic treatment after VTE assessment was defined from investigator's answer to the question "was the subject treated for VTE?" asked after diagnostic tests for suspected VTE and after lung imaging test for tumor evaluation.
Percentage of Participants Who Experienced Clinically Relevant Bleedings | From first study drug injection up to 3 days after last study drug injection
  Clinically Relevant Bleedings included overt bleedings classified by the CIAC as:
  * "major" (fatal, in a critical area/organ, causing a drop in hemoglobin ≥2 g/dL or requiring transfusion ≥2 units of blood)
  * "clinically relevant non-major" (requiring medical intervention and not meeting criteria for major bleeding).
Overall survival [OS] | From randomization up to 1 year after randomization or 7 months following randomization of the last participant, whichever came first
  Survival status was collected for all participants either one year after randomization, or at the study end date, (ie, 7 months following randomization of the last patient), whichever came first.
  OS was defined as the time from date of randomization to date of death due to any cause. Participants alive were censored at last date of contact that they were known to be alive.

OTHER OUTCOMES:
Platelets Count: Percentage of Participants With Potentially Clinically Significant Abnormalities [PCSA] | From first study drug injection up to 3 days after last study drug injection
  PCSA are abnormal values considered medically important by the Sponsor according to predefined criteria based on literature review.
  Thresholds for platelet counts were defined as follows:
  * Platelets count <50 Giga/L;
  * Platelets count ≥50 and <100 Giga/L;
Liver Function: Percentage of Participants With Potentially Clinically Significant Abnormalities [PCSA] | From first study drug injection up to 3 days after last study drug injection
  Thresholds were defined as follows:
  * Alanine Aminotransferase [ALAT] >3 Upper Normal Limit [ULN];
  * Total Bilirubin [TB] >2 ULN;
  * ALAT >3 ULN and TB >2 ULN;
  Cases with ALAT >3 ULN and TB >2 ULN (not necessarily concomitant) were evaluated by blinded independent adjudicator to determine if they met Hy's law criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Turpie, MD, Study Chair — HHS-General Hospital, Hamilton, Canada; Giancarlo Agnelli, MD, Principal Investigator — University Of Perugia
Locations (411):
- United States (48):
  - Investigational Site Number 840006, Birmingham, Alabama
  - Investigational Site Number 840007, Casa Grande, Arizona
  - Investigational Site Number 840060, Tucson, Arizona
  - Investigational Site Number 840050, Fountain Valley, California
  - Investigational Site Number 840072, Fullerton, California
  - Investigational Site Number 840037, Indian Wells, California
  - Investigational Site Number 840069, La Verne, California
  - Investigational Site Number 840009, Long Beach, California
  - Investigational Site Number 840001, Oceanside, California
  - Investigational Site Number 840011, Rancho Mirage, California
  - Investigational Site Number 840029, West Covina, California
  - Investigational Site Number 840005, Norwich, Connecticut
  - Investigational Site Number 840064, Torrington, Connecticut
  - Investigational Site Number 840038, Woodbridge, Connecticut
  - Investigational Site Number 840052, Washington D.C., District of Columbia
  - Investigational Site Number 840025, Washington D.C., District of Columbia
  - Investigational Site Number 840074, Clearwater, Florida
  - Investigational Site Number 840019, Jacksonville, Florida
  - Investigational Site Number 840051, Rockledge, Florida
  - Investigational Site Number 840073, Sarasota, Florida
  - Investigational Site Number 840070, Roswell, Georgia
  - Investigational Site Number 840016, Park Ridge, Illinois
  - Investigational Site Number 840028, Quincy, Illinois
  - Investigational Site Number 840008, Skokie, Illinois
  - Investigational Site Number 840033, Goshen, Indiana
  - Investigational Site Number 840010, Indianapolis, Indiana
  - Investigational Site Number 840014, Louisville, Kentucky
  - Investigational Site Number 840048, Mount Sterling, Kentucky
  - Investigational Site Number 840047, Metairie, Louisiana
  - Investigational Site Number 840032, Ruston, Louisiana
  - Investigational Site Number 840042, Bethesda, Maryland
  - Investigational Site Number 840066, Easton, Maryland
  - Investigational Site Number 840059, Tupelo, Mississippi
  - Investigational Site Number 840024, Rochester, New York
  - Investigational Site Number 840031, Syracuse, New York
  - Investigational Site Number 840020, Durham, North Carolina
  - Investigational Site Number 840021, Durham, North Carolina
  - Investigational Site Number 840026, High Point, North Carolina
  - Investigational Site Number 840046, Bismarck, North Dakota
  - Investigational Site Number 840003, Middletown, Ohio
  - Investigational Site Number 840022, Sylvania, Ohio
  - Investigational Site Number 840075, East Providence, Rhode Island
  - Investigational Site Number 840067, Beaumont, Texas
  - Investigational Site Number 840004, El Paso, Texas
  - Investigational Site Number 840034, Houston, Texas
  - Investigational Site Number 840035, Sugar Land, Texas
  - Investigational Site Number 840063, Kennewick, Washington
  - Investigational Site Number 840018, Tacoma, Washington
- Argentina (5):
  - Investigational Site Number 032006, Buenos Aires
  - Investigational Site Number 032003, Capital Federal
  - Investigational Site Number 032004, Rosario
  - Investigational Site Number 032007, San Miguel de Tucumán
  - Investigational Site Number 032005, San Miguel de Tucumán
- Australia (9):
  - Investigational Site Number 036004, Adelaide
  - Investigational Site Number 036002, Bedford Park
  - Investigational Site Number 036001, Box Hill
  - Investigational Site Number 036009, Lismore
  - Investigational Site Number 036007, Perth
  - Investigational Site Number 036006, Ringwood East
  - Investigational Site Number 036008, Westmead
  - Investigational Site Number 036003, Woodville
  - Investigational Site Number 036005, Woolloongabba
- Austria (3):
  - Investigational Site Number 040002, Graz
  - Investigational Site Number 040003, Vienna
  - Investigational Site Number 040004, Vienna
- Belarus (4):
  - Investigational Site Number 112002, Homyel
  - Investigational Site Number 112003, Minsk
  - Investigational Site Number 112001, Minsk
  - Investigational Site Number 112004, Vitebsk
- Belgium (10):
  - Investigational Site Number 056008, Bonheiden
  - Investigational Site Number 056011, Brussels
  - Investigational Site Number 056005, Ghent
  - Investigational Site Number 056010, Haine-Saint-Paul
  - Investigational Site Number 056006, Kortrijk
  - Investigational Site Number 056009, Liège
  - Investigational Site Number 056004, Merksem
  - Investigational Site Number 056003, Ostend
  - Investigational Site Number 056012, Ottignies
  - Investigational Site Number 056002, Sint-Niklaas
- Brazil (22):
  - Investigational Site Number 076002, Belo Horizonte
  - Investigational Site Number 076022, Curitiba
  - Investigational Site Number 076015, Curitiba
  - Investigational Site Number 076012, Florianópolis
  - Investigational Site Number 076001, Fortaleza
  - Investigational Site Number 076009, Goiânia
  - Investigational Site Number 076007, Goiânia
  - Investigational Site Number 076016, Goiânia
  - Investigational Site Number 076024, Ijuí
  - Investigational Site Number 076003, Joinville
  - Investigational Site Number 076010, Londrina
  - Investigational Site Number 076026, Passo Fundo
  - Investigational Site Number 076027, Passo Fundo
  - Investigational Site Number 076023, Porto Alegre
  - Investigational Site Number 076020, Porto Alegre
  - Investigational Site Number 076014, Salvador
  - Investigational Site Number 076018, Salvador
  - Investigational Site Number 076011, Santo André
  - Investigational Site Number 076006, São José dos Campos
  - Investigational Site Number 076008, São Paulo
  - Investigational Site Number 076017, São Paulo
  - Investigational Site Number 076004, Taguatinga
- Bulgaria (2):
  - Investigational Site Number 100001, Rousse
  - Investigational Site Number 100003, Varna
- Canada (11):
  - Investigational Site Number 124008, Greenfield Park
  - Investigational Site Number 124007, Kelowna
  - Investigational Site Number 124010, Moncton
  - Investigational Site Number 124003, Montreal
  - Investigational Site Number 124002, Ottawa
  - Investigational Site Number 124009, Owen Sound
  - Investigational Site Number 124006, Rimouski
  - Investigational Site Number 124013, Saint John
  - Investigational Site Number 124001, Sherbrooke
  - Investigational Site Number 124012, Victoria
  - Investigational Site Number 124011, Weston
- Investigational Site Number 152002, Temuco, Chile
- China (20):
  - Investigational Site Number 156014, Beijing
  - Investigational Site Number 156008, Beijing
  - Investigational Site Number 156022, Beijing
  - Investigational Site Number 156031, Changchun
  - Investigational Site Number 156021, Chengdu
  - Investigational Site Number 156019, Chongqing
  - Investigational Site Number 156003, Dalian
  - Investigational Site Number 156025, Guangzhou
  - Investigational Site Number 156026, Hangzhou
  - Investigational Site Number 156030, Nanning
  - Investigational Site Number 156029, Qingdao
  - Investigational Site Number 156024, Shanghai
  - Investigational Site Number 156028, Shanghai
  - Investigational Site Number 156020, Shanghai
  - Investigational Site Number 156011, Shanghai
  - Investigational Site Number 156013, Shantou
  - Investigational Site Number 156012, Suzhou
  - Investigational Site Number 156004, Xi'an
  - Investigational Site Number 156009, Xi'an
  - Investigational Site Number 156027, Yinchuan
- Colombia (7):
  - Investigational Site Number 170010, Bogotá
  - Investigational Site Number 170005, Manizales
  - Investigational Site Number 170002, Medellín
  - Investigational Site Number 170006, Medellín
  - Investigational Site Number 170007, Medellín
  - Investigational Site Number 170008, Montería
  - Investigational Site Number 170004, Pereira
- Croatia (7):
  - Investigational Site Number 191006, Pula
  - Investigational Site Number 191005, Rijeka
  - Investigational Site Number 191007, Varaždin
  - Investigational Site Number 191003, Zadar
  - Investigational Site Number 191008, Zagreb
  - Investigational Site Number 191001, Zagreb
  - Investigational Site Number 191004, Zagreb
- Czechia (4):
  - Investigational Site Number 203004, Hradec Králové
  - Investigational Site Number 203008, Kolín
  - Investigational Site Number 203007, Nová Ves pod Pleší
  - Investigational Site Number 203003, Prague
- Investigational Site Number 208001, Herlev, Denmark
- Investigational Site Number 233001, Tallinn, Estonia
- Investigational Site Number 246001, Turku, Finland
- France (16):
  - Investigational Site Number 250002, Antibes
  - Investigational Site Number 250010, Colmar
  - Investigational Site Number 250020, Gap
  - Investigational Site Number 250005, Lille
  - Investigational Site Number 250025, Lille
  - Investigational Site Number 250012, Lille
  - Investigational Site Number 250003, Lyon
  - Investigational Site Number 250001, Marseille
  - Investigational Site Number 250024, Montpellier
  - Investigational Site Number 250006, Paris
  - Investigational Site Number 250027, Paris
  - Investigational Site Number 250004, Paris
  - Investigational Site Number 250021, Reims
  - Investigational Site Number 250019, Rouen
  - Investigational Site Number 250017, Saint-Grégoire
  - Investigational Site Number 250014, Vandœuvre-lès-Nancy
- Germany (31):
  - Investigational Site Number 276012, Augsburg
  - Investigational Site Number 276025, Berlin
  - Investigational Site Number 276016, Berlin
  - Investigational Site Number 276002, Berlin
  - Investigational Site Number 276029, Berlin
  - Investigational Site Number 276004, Bochum
  - Investigational Site Number 276006, Cologne
  - Investigational Site Number 276014, Dresden
  - Investigational Site Number 276009, Dresden
  - Investigational Site Number 276030, Essen
  - Investigational Site Number 276005, Frankfurt am Main
  - Investigational Site Number 276032, Gauting
  - Investigational Site Number 276034, Halle
  - Investigational Site Number 276038, Halle
  - Investigational Site Number 276037, Hamburg
  - Investigational Site Number 276007, Hanover
  - Investigational Site Number 276020, Leer
  - Investigational Site Number 276010, Leipzig
  - Investigational Site Number 276017, Magdeburg
  - Investigational Site Number 276011, Mannheim
  - Investigational Site Number 276003, Minden
  - Investigational Site Number 276021, München
  - Investigational Site Number 276019, München
  - Investigational Site Number 276015, München
  - Investigational Site Number 276013, Neumünster
  - Investigational Site Number 276022, Oldenburg
  - Investigational Site Number 276035, Paderborn
  - Investigational Site Number 276031, Passau
  - Investigational Site Number 276023, Rosenheim
  - Investigational Site Number 276008, Singen
  - Investigational Site Number 276024, Westerstede
- Greece (3):
  - Investigational Site Number 300004, Athens
  - Investigational Site Number 300003, Heraklion
  - Investigational Site Number 300002, Thessaloniki
- Investigational Site Number 344001, Hong Kong, Hong Kong
- Hungary (11):
  - Investigational Site Number 348005, Budapest
  - Investigational Site Number 348006, Budapest
  - Investigational Site Number 348009, Budapest
  - Investigational Site Number 348004, Budapest
  - Investigational Site Number 348010, Farkasgyepű
  - Investigational Site Number 348001, Gyula
  - Investigational Site Number 348012, Mátraháza
  - Investigational Site Number 348003, Sopron
  - Investigational Site Number 348008, Szikszó
  - Investigational Site Number 348011, Szolnok
  - Investigational Site Number 348007, Zalaegerszeg
- India (21):
  - Investigational Site Number 356006, Bangalore
  - Investigational Site Number 356008, Bangalore
  - Investigational Site Number 356009, Bhopal
  - Investigational Site Number 356018, Chennai
  - Investigational Site Number 356020, Chennai
  - Investigational Site Number 356019, Coimbatore
  - Investigational Site Number 356015, Hyderabad
  - Investigational Site Number 356025, Hyderabad
  - Investigational Site Number 356011, Jaipur
  - Investigational Site Number 356014, Kochi
  - Investigational Site Number 356003, Kolkata
  - Investigational Site Number 356013, Kolkata
  - Investigational Site Number 356017, Kolkata
  - Investigational Site Number 356005, Madurai
  - Investigational Site Number 356016, Miraj
  - Investigational Site Number 356001, Mumbai
  - Investigational Site Number 356023, Nagpur
  - Investigational Site Number 356002, New Delhi
  - Investigational Site Number 356004, Pune
  - Investigational Site Number 356024, Pune
  - Investigational Site Number 356012, Visakhapatnam
- Indonesia (3):
  - Investigational Site Number 360002, Bandung
  - Investigational Site Number 360001, Denpasar
  - Investigational Site Number 360004, Medan
- Ireland (3):
  - Investigational Site Number 372003, Dublin
  - Investigational Site Number 372002, Dublin
  - Investigational Site Number 372004, Dublin
- Israel (5):
  - Investigational Site Number 376003, Jerusalem
  - Investigational Site Number 376004, Kfar Saba
  - Investigational Site Number 376001, Nahariya
  - Investigational Site Number 376006, Petah Tikva
  - Investigational Site Number 376007, Tzrifin
- Italy (18):
  - Investigational Site Number 380005, Castellanza
  - Investigational Site Number 380014, Cattolica
  - Investigational Site Number 380007, Cesena
  - Investigational Site Number 380015, Cremona
  - Investigational Site Number 380009, Faenza
  - Investigational Site Number 380012, Lecce
  - Investigational Site Number 380006, Lugo
  - Investigational Site Number 380001, Meldola
  - Investigational Site Number 380011, Parma
  - Investigational Site Number 380020, Perugia
  - Investigational Site Number 380013, Ravenna
  - Investigational Site Number 380016, Rimini
  - Investigational Site Number 380004, Sondrio
  - Investigational Site Number 380010, Sora
  - Investigational Site Number 380008, Taormina
  - Investigational Site Number 380019, Terni
  - Investigational Site Number 380003, Treviglio
  - Investigational Site Number 380017, Udine
- Latvia (3):
  - Investigational Site Number 428002, Liepāja
  - Investigational Site Number 428003, Riga
  - Investigational Site Number 428001, Riga
- Lithuania (2):
  - Investigational Site Number 440001, Kaunas
  - Investigational Site Number 440002, Vilnius
- Malaysia (4):
  - Investigational Site Number 458004, George Town
  - Investigational Site Number 458005, George Town
  - Investigational Site Number 458001, Kota Kinabalu
  - Investigational Site Number 458003, Kuala Lumpur
- Mexico (7):
  - Investigational Site Number 484002, Acapulco
  - Investigational Site Number 484006, Aguascalientes
  - Investigational Site Number 484007, Durango
  - Investigational Site Number 484008, Mérida
  - Investigational Site Number 484012, Puebla City
  - Investigational Site Number 484003, Toluca
  - Investigational Site Number 484010, Xalapa
- Netherlands (5):
  - Investigational Site Number 528004, Groningen
  - Investigational Site Number 528005, Helmond
  - Investigational Site Number 528001, Hoofddorp
  - Investigational Site Number 528003, Rotterdam
  - Investigational Site Number 528006, The Hague
- Investigational Site Number 578001, Oslo, Norway
- Peru (12):
  - Investigational Site Number 604012, Arequipa
  - Investigational Site Number 604004, Callao
  - Investigational Site Number 604011, Callao
  - Investigational Site Number 604001, Cercado
  - Investigational Site Number 604002, Chiclayo
  - Investigational Site Number 604008, Lima
  - Investigational Site Number 604007, Lima
  - Investigational Site Number 604009, Lima
  - Investigational Site Number 604005, Lima
  - Investigational Site Number 604006, Lima
  - Investigational Site Number 604010, Lima
  - Investigational Site Number 604003, Lima
- Poland (15):
  - Investigational Site Number 616009, Bialystok
  - Investigational Site Number 616008, Bielsko-Biala
  - Investigational Site Number 616006, Gliwice
  - Investigational Site Number 616004, Krakow
  - Investigational Site Number 616003, Lubin
  - Investigational Site Number 616019, Olsztyn
  - Investigational Site Number 616021, Otwock
  - Investigational Site Number 616010, Poznan
  - Investigational Site Number 616001, Prabuty
  - Investigational Site Number 616014, Rybnik
  - Investigational Site Number 616005, Rzeszów
  - Investigational Site Number 616013, Torun
  - Investigational Site Number 616018, Warsaw
  - Investigational Site Number 616002, Warsaw
  - Investigational Site Number 616015, Wroclaw
- Portugal (6):
  - Investigational Site Number 620003, Aveiro
  - Investigational Site Number 620009, Guimarães
  - Investigational Site Number 620004, Lisbon
  - Investigational Site Number 620008, Matosinhos Municipality
  - Investigational Site Number 620007, Porto
  - Investigational Site Number 620002, Setúbal
- Romania (7):
  - Investigational Site Number 642004, Brasov
  - Investigational Site Number 642002, Bucharest
  - Investigational Site Number 642001, Cluj-Napoca
  - Investigational Site Number 642006, Cluj-Napoca
  - Investigational Site Number 642010, Iași
  - Investigational Site Number 642003, Suceava
  - Investigational Site Number 642008, Timișoara
- Russia (22):
  - Investigational Site Number 643024, Berdsk
  - Investigational Site Number 643006, Chelyabinsk
  - Investigational Site Number 643001, Kazan'
  - Investigational Site Number 643004, Krasnoyarsk
  - Investigational Site Number 643010, Obninsk
  - Investigational Site Number 643005, Omsk
  - Investigational Site Number 643022, Pyatigorsk
  - Investigational Site Number 643023, Rostov-on-Don
  - Investigational Site Number 643009, Saint Petersburg
  - Investigational Site Number 643014, Saint Petersburg
  - Investigational Site Number 643015, Saint Petersburg
  - Investigational Site Number 643011, Saint Petersburg
  - Investigational Site Number 643020, Saratov
  - Investigational Site Number 643019, Smolensk
  - Investigational Site Number 643021, Sochi
  - Investigational Site Number 643008, Tomsk
  - Investigational Site Number 643016, Tula
  - Investigational Site Number 643018, Tyumen
  - Investigational Site Number 643012, Ufa
  - Investigational Site Number 643007, Vladivostok
  - Investigational Site Number 643017, Voronezh
  - Investigational Site Number 643003, Yaroslavl
- Serbia (4):
  - Investigational Site Number 688002, Belgrade
  - Investigational Site Number 688004, Belgrade
  - Investigational Site Number 688007, Kragujevac
  - Investigational Site Number 688005, Niš
- Investigational Site Number 703003, Trnava, Slovakia
- Slovenia (2):
  - Investigational Site Number 705003, Golnik
  - Investigational Site Number 705002, Maribor
- South Africa (2):
  - Investigational Site Number 710003, Durban
  - Investigational Site Number 710002, Durban
- South Korea (9):
  - Investigational Site Number 410008, Daegu
  - Investigational Site Number 410007, Seoul
  - Investigational Site Number 410001, Seoul
  - Investigational Site Number 410002, Seoul
  - Investigational Site Number 410006, Seoul
  - Investigational Site Number 410005, Seoul
  - Investigational Site Number 410003, Seoul
  - Investigational Site Number 410009, Seoul
  - Investigational Site Number 410004, Suwon
- Spain (12):
  - Investigational Site Number 724008, Barakaldo
  - Investigational Site Number 724010, Barakaldo
  - Investigational Site Number 724004, Barcelona
  - Investigational Site Number 724006, Islas Baleares
  - Investigational Site Number 724011, Lleida
  - Investigational Site Number 724001, Madrid
  - Investigational Site Number 724007, Madrid
  - Investigational Site Number 724013, Madrid
  - Investigational Site Number 724012, Madrid
  - Investigational Site Number 724005, Ourense
  - Investigational Site Number 724003, Port de Sagunt
  - Investigational Site Number 724002, Valencia
- Sweden (4):
  - Investigational Site Number 752003, Gothenburg
  - Investigational Site Number 752005, Mora
  - Investigational Site Number 752002, Uppsala
  - Investigational Site Number 752001, Vaxjo
- Switzerland (2):
  - Investigational Site Number 756006, Aarau
  - Investigational Site Number 756004, Winterthur
- Investigational Site Number 158004, Changhua, Taiwan
- Ukraine (9):
  - Investigational Site Number 804008, Cherkasy
  - Investigational Site Number 804009, Chernivtsi
  - Investigational Site Number 804002, Dnipropetrovsk
  - Investigational Site Number 804006, Donetsk
  - Investigational Site Number 804005, Kryvyi Rih
  - Investigational Site Number 804001, Lutsk
  - Investigational Site Number 804010, Lviv
  - Investigational Site Number 804011, Sumy
  - Investigational Site Number 804004, Ternopil
- United Kingdom (13):
  - Investigational Site Number 826016, Bangor
  - Investigational Site Number 826010, Brighton
  - Investigational Site Number 826015, Coventry
  - Investigational Site Number 826013, Dundee
  - Investigational Site Number 826007, Hull
  - Investigational Site Number 826002, Lincoln
  - Investigational Site Number 826017, Lincoln
  - Investigational Site Number 826005, Manchester
  - Investigational Site Number 826014, Metropolitan Borough of Wirral
  - Investigational Site Number 826004, Norwich
  - Investigational Site Number 826009, Peterborough
  - Investigational Site Number 826011, Portsmouth
  - Investigational Site Number 826001, Shrewsbury

REFERENCES:
- [Result] Agnelli G, George DJ, Kakkar AK, Fisher W, Lassen MR, Mismetti P, Mouret P, Chaudhari U, Lawson F, Turpie AG; SAVE-ONCO Investigators. Semuloparin for thromboprophylaxis in patients receiving chemotherapy for cancer. N Engl J Med. 2012 Feb 16;366(7):601-9. doi: 10.1056/NEJMoa1108898. PMID 22335737
- [Derived] Rutjes AW, Porreca E, Candeloro M, Valeriani E, Di Nisio M. Primary prophylaxis for venous thromboembolism in ambulatory cancer patients receiving chemotherapy. Cochrane Database Syst Rev. 2020 Dec 18;12(12):CD008500. doi: 10.1002/14651858.CD008500.pub5. PMID 33337539